CLINICAL TRIAL: NCT02408302
Title: Buccal Midazolam Versus Nasal or Oral Midazolam Sedation for Minor Invasive Procedures in Children: A Prospective Randomized Control Study
Brief Title: Buccal Midazolam Versus Nasal or Oral Midazolam Sedation for Minor Invasive Procedures in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Muriel Konopnicki, Head of Pediatric emergency room, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CMC-13-0075-CTIL
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Dormicum; Conscious Sedation; Children
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- oral midazolam (Active Comparator): oral midazolam 0.5-0.7 mg/kg maximum 10 mg. one dose only before the invasive procedure.
  Interventions: Drug: Midazolam
- intranasal midazolam (Active Comparator): intranasal midazolam 0.3-0.5 mg/kg maximum 5 mg. one dose only before the invasive procedure
  Interventions: Drug: Midazolam
- buccal midazolam (Active Comparator): buccal midazolam 0.3-0.5 mg/kg maximum 5 mg. one dose only before the invasive procedure
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — comparison between 3 routes of administration of the drug Midazolam used for sedation for minor procedures in pediatric population. the routes are oral intranasal and buccal.
  Other Names: Dormicum

SUMMARY:
Currently Midazolam sedation is the standard of care for minor invasive procedures in pediatric patients; its use is restricted to two routes of administration for this purpose oral and intranasal.

A third route of administration (buccal) is tested and approved for seizure management. In the investigators' study the researchers investigate the buccal route of administration versus oral or intranasal administration for sedation. The investigators' hypothesis is that buccal route of administration is more convenient than intranasal and better absorbed than oral.

ELIGIBILITY:
Inclusion Criteria:

* age 5 months to 6 years.
* need to undergo a minimal invasive procedure that requires light sedation.
* ASA (American Society of Anesthesiologists) I-II
* parent that can read, understand and sign an informed consent form

Exclusion Criteria:

* patients with life threatening conditions.
* patients with respiratory or cardiac chronic illnesses or ASA other than I-II.
* patients with traumatic injury for the nose or the oral cavity.
* patients that would not or cannot take the drug in the route picked in a randomized way.

Ages: 5 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
time until sedation is achieved | 1 hour
duration of sedation | 4 hour
  time from achieving sedation until reaching full consciousness
convenience of administration | 15 minutes
  described by the parent and the physician by a numerical rating scale (NRS) questionaire
efficacy of the sedation | 4 hours
  described by the parent, nurse and physician by a NRS questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Konopnicki, Principal Investigator — Carmal Medical Center, Haifa, Israel
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Krauss B, Green SM. Sedation and analgesia for procedures in children. N Engl J Med. 2000 Mar 30;342(13):938-45. doi: 10.1056/NEJM200003303421306. No abstract available. PMID 10738053
- [Background] Krauss B, Green SM. Procedural sedation and analgesia in children. Lancet. 2006 Mar 4;367(9512):766-80. doi: 10.1016/S0140-6736(06)68230-5. PMID 16517277
- [Background] American Academy of Pediatrics; American Academy of Pediatric Dentistry; Cote CJ, Wilson S; Work Group on Sedation. Guidelines for monitoring and management of pediatric patients during and after sedation for diagnostic and therapeutic procedures: an update. Pediatrics. 2006 Dec;118(6):2587-602. doi: 10.1542/peds.2006-2780. PMID 17142550
- [Background] Procacci P, Francini F, Zoppi M, Maresca M. Cutaneous pain threshold changes after sympathetic block in reflex dystrophies. Pain. 1975 Jun;1(2):167-175. doi: 10.1016/0304-3959(75)90100-1. PMID 1235980
- [Background] American Society of Anesthesiologists Task Force on Sedation and Analgesia by Non-Anesthesiologists. Practice guidelines for sedation and analgesia by non-anesthesiologists. Anesthesiology. 2002 Apr;96(4):1004-17. doi: 10.1097/00000542-200204000-00031. No abstract available. PMID 11964611
- [Background] Godwin SA, Caro DA, Wolf SJ, Jagoda AS, Charles R, Marett BE, Moore J; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2005 Feb;45(2):177-96. doi: 10.1016/j.annemergmed.2004.11.002. No abstract available. PMID 15671976
- [Background] Shavit I, Feraru L, Miron D, Weiser G. Midazolam for urethral catheterisation in female infants with suspected urinary tract infection: a case-control study. Emerg Med J. 2014 Apr;31(4):278-80. doi: 10.1136/emermed-2012-202088. Epub 2013 Feb 22. PMID 23435653
- [Background] McErlean M, Bartfield JM, Karunakar TA, Whitman MC, Turley DM. Midazolam syrup as a premedication to reduce the discomfort associated with pediatric intravenous catheter insertion. J Pediatr. 2003 Apr;142(4):429-30. doi: 10.1067/mpd.2003.62. PMID 12712062
- [Background] Lane RD, Schunk JE. Atomized intranasal midazolam use for minor procedures in the pediatric emergency department. Pediatr Emerg Care. 2008 May;24(5):300-3. doi: 10.1097/PEC.0b013e31816ecb6f. PMID 18496113
- [Background] Wiznitzer M. Buccal midazolam is effective for acute treatment of seizures. J Pediatr. 2006 Jan;148(1):143. doi: 10.1016/j.jpeds.2005.12.008. No abstract available. PMID 16440479
- [Background] Wiznitzer M. Buccal midazolam for seizures. Lancet. 2005 Jul 16-22;366(9481):182-3. doi: 10.1016/S0140-6736(05)66884-5. No abstract available. PMID 16023491